CLINICAL TRIAL: NCT00310700
Title: A Phase IV, Single Centre, Open-label Study to Investigate the Kinetics of the B Cell Response to the First and the Third Immunization With Chiron Meningococcal C Conjugate Vaccine Administered to Healthy Infants at 2, 3 and 4 Months of Age
Brief Title: Kinetics of B Cell Response in Infants Menjugate Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M14P5; Impact N° 1457; 2004-004962-33 (EudraCT Number)
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; vaccines, conjugate; immunology; infant; antibody persistence
MeSH Terms: interventions — serogroup C meningococcal conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C conjugate vaccine

SUMMARY:
Kinetics of B cell response in infants Menjugate vaccination

ELIGIBILITY:
Inclusion Criteria:

* healthy infants

Exclusion Criteria:

* previously ascertained or suspected disease caused by N. meningitidis
* previous household contact with an individual with a positive culture of N. meningitidis serogroup C

Ages: 8 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To establish at which day meningococcal C specific B cells are detectable in the blood of healthy infants following first and third immunisation with MenC Conjugate Vaccine as determined by Men C specific B-cell ELISPot assay.

SECONDARY OUTCOMES:
To establish how long the B cells persist in the blood
To note the difference between plasma cell response following the first and third MenC vaccination.
To determine the immune response to Neisseria meningitidis serogroup C 26-34 days after the third immunisation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, Oxon, United Kingdom

REFERENCES:
- [Background] Kelly DF, Snape MD, Perrett KP, Clutterbuck EA, Lewis S, Blanchard Rohner G, Jones M, Yu LM, Pollard AJ. Plasma and memory B-cell kinetics in infants following a primary schedule of CRM 197-conjugated serogroup C meningococcal polysaccharide vaccine. Immunology. 2009 May;127(1):134-43. doi: 10.1111/j.1365-2567.2008.02934.x. PMID 19175802